CLINICAL TRIAL: NCT02163616
Title: Treatment of Postpartum Hemorrhage With Misoprostol: Who do we Treat? Who Will Develop Fever?
Brief Title: Treatment of Postpartum Hemorrhage With Misoprostol: Fever Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Centro Rosarino de Estudios Perinatales (Unknown); University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3003
Record Dates: First submitted 2014-06-06; First posted 2014-06-13 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Postpartum Hemorrhage
Keywords: Primary postpartum hemorrhage; PPH; uterine atony; high fever; hyperpyrexia; shock index
MeSH Terms: conditions — Postpartum Hemorrhage; Uterine Inertia; Hyperthermia | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PPH Treatment (Experimental): 800mcg sublingual misoprostol
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — 800 mcg of sublingual misoprostol

SUMMARY:
This study seeks to assess whether populations of women in Latin America outside Quito, Ecuador are at increased risk for developing elevated body temperature above 40.0°C following PPH treatment with 800mcg sublingual misoprostol. The study will be carried out in hospitals representative of different regions of Latin America to explore environmental and genetic hypotheses related to the occurrence of misoprostol-induced fever. Postpartum blood loss, pulse and blood pressure will be systematically measured for all women enrolled to explore new clinical indicators for identifying women who require clinical intervention for excessive bleeding. Blood samples will be collected among women treated with misoprostol to investigate genetic factors responsible for elevated body temperature induced by misoprostol.

The investigators hypothesize that rates of high fever (≥40.0°C) following misoprostol treatment (800mcg given sublingually) will be variable across settings. The investigators expect that the side effect profile following 800 mcg misoprostol given sublingually, in particular the rates of any shivering and fever ≥38.0°C, will be comparable to previous results using misoprostol for PPH.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give informed consent
* Vaginal delivery
* Postpartum hemorrhage due to suspected uterine atony
* Able and willing to give informed consent

Exclusion Criteria:

* Known allergy to misoprostol or other prostaglandins
* Underwent a c-section during the current delivery
* Unable to provide informed consent due to mental impairment, distress during labor or other reason
* Unwilling and/or unable to respond to brief questionnaires or have her blood drawn

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 635 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Rates of high fever (≥40.0°C) | First 2 hours postpartum
  Percentage of women with body temperature measures ≥40°C

SECONDARY OUTCOMES:
Side effect profile of misoprostol for PPH treatment | Side effects observed for 3 hours post-treatment with misoprostol for PPH
  Percentage of women experiencing any shivering and any fever or any other side effect
Acceptability of regimen and side effects to women | Interviewed prior to hospital discharge (about 24 hours postpartum)
  Percentage of women who rate side effects as acceptable, neutral, unacceptable, don't know
Shock index values | First hour of the puerperium
  Pulse and blood pressure will be measured at pre-defined intervals (15, 30, 45, and 60 minutes)
Genetic factors responsible for elevated body temperature | sample taken 24-48 hours postpartum
  Blood samples will be collected among women enrolled and sent to the Wolfson centre for personalized medicine at the University of Liverpool for genetic analysis to investigate genetic markers associated with misoprostol-induced fever.

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects; Guillermo Carroli, MD, Principal Investigator — Centro Rosarino de Estudios Perinatales; Jill Durocher, Principal Investigator — Gynuity Health Projects; Ilana Dzuba, MPH, Principal Investigator — Gynuity Health Projects
Locations (2):
- Argentina (2):
  - Hospital Dr. A. Llano, Corrientes
  - Hospital J.R. Vidal, Corrientes

REFERENCES:
- See also: Gynuity Health Projects — http://www.gynuity.org